CLINICAL TRIAL: NCT05419492
Title: ENDEAVOR: A Clinical Study to Evaluate the Safety and Efficacy of ETX101, an AAV9-Delivered Gene Therapy in Infants and Children With SCN1A-Positive Dravet Syndrome
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of ETX101 in Infants and Children With SCN1A-Positive Dravet Syndrome
Acronym: ENDEAVOR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Encoded Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETX-DS-002
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-01

CONDITIONS: Dravet Syndrome
Keywords: Dravet; SCN1A; DEE; developmental and epileptic encephalopathy; Dravet Syndrome; SCN1A-positive; SCN1A+
MeSH Terms: conditions — Epilepsies, Myoclonic; Generalized Epilepsy With Febrile Seizures Plus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is open-label with no blinding.
  Part 2 will be conducted in a double-blinded manner whereby all Primary Site Staff (including clinicians, research coordinators, neuropsychologists, pharmacists, and physical therapists), study participants and caregivers, Sponsor and Sponsor-designees will be blinded through the end of Week 52 following Day 1 for each participant. The Surgical Site Staff will be unblinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (Experimental): Part 1 will follow an open-label, rule-based, dose-escalation design and will evaluate up to 4 dose levels of ETX101.
  Interventions: Drug: ETX101
- Part 2 (Sham Comparator): Part 2 is a dose-selection study, which will follow a double-blind (up through Week 52), randomized, sham delayed-treatment control design.
  There will be up to 3 cohorts in Part 2. If it is determined two dose levels of ETX101 will be evaluated in Part 2, participants will be randomized 1:1:1 to study treatment or sham procedure with delayed treatment. If Part 2 proceeds with a single dose level of ETX101, participants will be randomized 2:1 to study treatment or sham procedure with delayed treatment.
  Interventions: Drug: ETX101

INTERVENTIONS:
Drug: ETX101 — ETX101 is a non-replicating, recombinant adeno-associated viral vector serotype 9 (rAAV9) comprising a GABAergic regulatory element (reGABA) and an engineered transcription factor that increases transcription of the SCN1A gene (eTFSCN1A). ETX101 is intended as a one-time intracerebroventricular (ICV) administration.

SUMMARY:
ENDEAVOR is a Phase 1/2, 2-part, multicenter study to evaluate the safety and efficacy of ETX101 in participants with SCN1A-positive Dravet syndrome aged ≥6 to <36 months (Part 1) and aged ≥6 to <48 months (Part 2). Part 1 follows an open-label, dose-escalation design, and Part 2 is a randomized, double-blind, sham delayed-treatment control, dose-selection study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged between ≥6 months and <36 months in Part 1 and <48 months in Part 2.
* Participant must have a predicted loss of function pathogenic or likely pathogenic SCN1A variant.
* Participant must have experienced their first seizure between the ages of 3 and 15 months.
* Participant must have a clinical diagnosis of Dravet syndrome or the treating clinician must have a high clinical suspicion of a diagnosis of Dravet syndrome.
* Participant is receiving at least one prophylactic antiseizure medication.

Exclusion Criteria:

* Participant has another genetic mutation or clinical comorbidity which could potentially confound the typical Dravet phenotype.
* Participant has a known central nervous system structural and/or vascular abnormality (indicated by an MRI or CT scan of the brain).
* Participant has an abnormality that may interfere with CSF distribution and/or has an existing ventriculoperitoneal shunt.
* Participant is currently taking or has taken antiseizure medications (ASMs) at a therapeutic dose that are contraindicated in Dravet syndrome, including sodium channel blockers.
* Participant has experienced seizure freedom for a period of 4 consecutive weeks within the 90-day period prior to informed consent.
* Participant has previously received gene or cell therapy.
* Participant is currently enrolled in a clinical trial or receiving an investigational therapy, including under an expanded access and/or compassionate use program.
* Participant has clinically significant underlying liver disease.

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Proportions of participants experiencing any treatment-emergent adverse events (AEs), serious adverse events (SAEs), related AEs, AEs with severity Grade ≥ 3, AEs resulting in study discontinuation, and AEs with a fatal outcome. | Day 1 through Study Completion
Percent change in monthly countable seizure frequency (MCSF) period, with countable seizures defined as generalized tonic-clonic/clonic, focal motor with clearly observable clinical signs, tonic, or atonic seizures. | Between the pre-dose period (Part 1: 30 days prior to consent and the collection period through Day -1; Part 2: collection period between Day -72 and Day -1) and the 48-week post dosing period (defined as Week 5 through Week 52)

SECONDARY OUTCOMES:
Absolute change in monthly countable seizure frequency (MCSF) | Between the pre-dose period (Part 1: 30 days prior to consent and the collection period through Day -1; Part 2: collection period between Day -72 and Day -1) and the 48-week post dosing period (defined as Week 5 through Week 52)
Proportion of participants with ≥ 90% reduction in monthly countable seizure frequency (MCSF). | Between the pre-dose period (Part 1: 30 days prior to consent and the collection period through Day -1; Part 2: collection period between Day -72 and Day -1) and the 48-week post dosing period (defined as Week 5 through Week 52)
Change from baseline in the Vineland-3 Expressive Communication raw score at Week 52 | Baseline through Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Rico, M.D., Ph.D, Study Director — Encoded Therapeutics
Locations (3):
- United States (3):
  - UCSF Benioff Children's Hospitals, San Francisco, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No